CLINICAL TRIAL: NCT03962322
Title: Diaphragmatic Tissue Doppler During Weaning From Mechanical Ventilation
Acronym: TDD-wean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Principal Investigator, MD of ICU staff, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 23/19
Record Dates: First submitted 2019-05-13; First posted 2019-05-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: Diaphragmatic Tissue Doppler; Weaning; Mechanical ventilation

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weaning TDI (Experimental): A tissue doppler evaluation, using a sector transducer, will be performed by analyzing the diaphragmatic displacement velocity during inspiration and expiration in the modality of ventilation which precedes the trial, during the SBT and after extubation.
  Interventions: Other: Weaning TDI

INTERVENTIONS:
Other: Weaning TDI — Patients will be subjected to a spontaneous breathing test (Cpap 5), that consists in applying a positive end-expiratory pressure of 5 cm H2O for 20 minutes.
  A tissue doppler evaluation will then be performed by analyzing the diaphragmatic displacement velocity during inspiration and expiration and calculating the speed of muscles displacement and other derived index of muscle function in the modality of ventilation which precedes the trial, during the SBT and after extubation.

SUMMARY:
Weaning from mechanical ventilation is a critical issue and the diaphragmatic disfunction has been demonstrated to play an important role in extubation failure. the aim of present investigation is to evaluate diaphragmatic excursion velocity during in patients undergoing spontaneous breathing trial through tissue Doppler analysis in both inspiration and expiration.

DETAILED DESCRIPTION:
Tobin Index (RSBI), which is the ratio between respiratory rate (RR) and tidal volume (VT), is one of the most used indices to predict weaning outcome. The diaphragm plays a key role in generating VT and, in the case of diaphragmatic dysfunction, inspiratory accessory muscles may contribute to support ventilation. If this occurs during a spontaneous breathing trial (SBT), it will probably result in delayed weaning, since the accessory muscles are more fatigable than the diaphragm.

The diaphragmatic tissue Doppler imaging (TDI) is an ultrasonographic technique derived from ultrasound evaluation of heart's motility. Being a muscle doppler assessment, it can be easily used on the diaphragm to calculate the speed of muscles displacement that could be associated with patient's respiratory drive, as well as other derived index of muscle function.

The aim of the study is to measure the variations of diaphragmatic displacement velocities before and during the spontaneous breathing trial, useful to check if the patient is ready to breathe spontaneously. An observational study will be performed. Patients who are ready to be weaned will be subjected to a spontaneous breathing test (Cpap 5), that consists of applying a positive end-expiratory pressure of 5 cm H2O for 20 minutes. A tissue Doppler evaluation will then be performed by analyzing the diaphragmatic displacement velocity during inspiration and expiration in the modality of ventilation which precedes the trial and during the SBT.

Vital parameters will be monitored during the study. Mechanical ventilation length, incidence of tracheostomies, ICU and hospital recovery duration and hospital mortality will also be acquired.

ELIGIBILITY:
Inclusion Criteria:

* mechanical invasive ventilation ≥ 24 h
* readiness for extubation

Exclusion Criteria:

* refusal to grant consent
* pregnancy
* hemodynamic instability
* difficult management of secretions
* request for inotropy and/or vasoactive drugs at high doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure - Change in diaphragmatic displacement velocity | through each trial completion, an average of 20 minutes
  Inspiratory and expiratory diaphragmatic displacement velocity evaluated with tissue doppler during the assisted ventilation modality which preceded the trial, during the spontaneous breathing trial ( CPAP 5 ) and in spontaneous breathing.

SECONDARY OUTCOMES:
Diaphragmatic acceleration and deceleration | through each trial completion, an average of 20 minutes
  Diaphragmatic acceleration and deceleration evaluated with tissue doppler during the assisted ventilation modality which preceded the trial, during the spontaneous breathing trial ( CPAP 5 ) and in spontaneous breathing.
Gas exchange - arterial carbon dioxide tension | through each trial completion, an average of 20 minutes
  Arterial blood gases sample
Gas exchange - pH | through each trial completion, an average of 20 minutes
  Arterial blood gases sample
Gas exchange - arterial oxygen tension | through each trial completion, an average of 20 min
  Arterial blood gases sample
Dyspnea level | through each trial completion, an average of 20 minutes
  Dyspnea level will be evaluated through visual analogical scale ( VAS dyspnea). The dyspnea visual analog scale is represented by a 20 cm horizontal line. The ends are defined as the extreme limits of dyspnea from the left-lower end best, "not at all breathless"-to the right-upper end worst, "extremely breathless". Subjects will be instructed to indicate on the line the point corresponding to their breathlessness perception.
Heart rate | through each trial completion, an average of 20 minutes
  Heart Rate (HR) averages during each of the 3 ventilatory modes
Number of patients who experienced weaning failure | over 48 hours following extubation
  the need for non invasive ventilation or re-intubation due to any cause
Blood Pressure | through each trial completion, an average of 20 minutes
  Mean arterial Blood Pressure (BP) averages during each of the 3 ventilatory modes

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobin MJ. Respiratory monitoring in the intensive care unit. Am Rev Respir Dis. 1988 Dec;138(6):1625-42. doi: 10.1164/ajrccm/138.6.1625. PMID 3144222
- [Derived] Cammarota G, Boniolo E, Santangelo E, De Vita N, Verdina F, Crudo S, Sguazzotti I, Perucca R, Messina A, Zanoni M, Azzolina D, Navalesi P, Longhini F, Vetrugno L, Bignami E, Della Corte F, Tarquini R, De Robertis E, Vaschetto R. Diaphragmatic Kinetics Assessment by Tissue Doppler Imaging and Extubation Outcome. Respir Care. 2021 Jun;66(6):983-993. doi: 10.4187/respcare.08702. Epub 2021 Apr 27. PMID 33906957